CLINICAL TRIAL: NCT04430738
Title: A Phase 1b/2 Dose Escalation and Expansion Study of Tucatinib in Combination With Trastuzumab and Oxaliplatin-based Chemotherapy or Pembrolizumab-containing Combinations for HER2+ Gastrointestinal Cancers
Brief Title: Tucatinib Plus Trastuzumab and Oxaliplatin-based Chemotherapy or Pembrolizumab-containing Combinations for HER2+ Gastrointestinal Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-024; C4251005 (Other: Alias Study Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Carcinoma; Gastric Adenocarcinoma; GEJ Adenocarcinoma; Esophageal Adenocarcinoma; Cholangiocarcinoma; Gallbladder Carcinoma
Keywords: HER2+; HER2-positive; CRC; Gastric cancer; Esophageal cancer; Seattle Genetics
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma Of Esophagus; Cholangiocarcinoma; Gallbladder Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — tucatinib; Trastuzumab; Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1A (Experimental): Tucatinib + trastuzumab + FOLFOX given in 14-day cycles
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil
- Cohort 1B (Experimental): Tucatinib + trastuzumab + FOLFOX given in 14-day cycles
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil
- Cohort 1C (Experimental): Tucatinib + trastuzumab + CAPOX given in 21-day cycles
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: capecitabine
- Cohort 1D (Experimental): Tucatinib + trastuzumab + FOLFOX. Tucatinib and FOLFOX given in 14-day cycles and trastuzumab given every 21 days
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil
- Cohort 1E (Experimental): Tucatinib + trastuzumab + pembrolizumab + FOLFOX. Tucatinib and FOLFOX given in 14-day cycles, trastuzumab given in 21-day cycles, and pembrolizumab given in 42-day cycles
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Drug: pembrolizumab
- Cohort 1F (Experimental): Tucatinib + trastuzumab + pembrolizumab + CAPOX. Tucatinib, trastuzumab, and CAPOX given in 21-day cycles and pembrolizumab given in 42-day cycles.
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: capecitabine; Drug: pembrolizumab
- Cohort 1G (Experimental): Tucatinib + trastuzumab + pembrolizumab. Tucatinib and trastuzumab given in 21-day cycles and pembrolizumab given in 42-day cycles.
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: pembrolizumab
- Cohort 2A (Experimental): Tucatinib + trastuzumab + pembrolizumab + (FOLFOX or CAPOX). Either (1) tucatinib and FOLFOX given in 14-day cycles or (2) tucatinib and CAPOX given in 21-day cycles. Trastuzumab given in 21-day cycles and pembrolizumab given in 42-day cycles.
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Drug: capecitabine; Drug: pembrolizumab
- Cohort 2B (Experimental): Tucatinib + trastuzumab + FOLFOX given in 14-day cycles.
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil

INTERVENTIONS:
Drug: tucatinib — For Cohort 1A, 150 mg will be administered twice daily by mouth (orally) from Cycle 1 Day 8 onwards. For all other cohorts, 300 mg (or intermediate dose) will be given orally twice daily starting on Cycle 1 Day 1.
  Other Names: TUKYSA
Drug: trastuzumab — Cohorts 1A and 1B: a 6 mg/kg loading dose will be given into the vein (IV; intravenously) on Cycle 1 Day 1, followed by a dose of 4 mg/kg IV every 2 weeks starting on Cycle 2 Day 1. Cohorts 1C, 1D, 1E, 1F, 1G, 2A, and 2B: an 8 mg/kg loading dose will be administered IV on Cycle 1 Day 1, followed by a dose of 6 mg/kg IV every 3 weeks thereafter.
Drug: oxaliplatin — 85 mg/m^2 given IV every 2 weeks for cohorts using FOLFOX. For cohorts using CAPOX regimen, 130 mg/m^2 given every 3 weeks.
  Arms: Cohort 1A; Cohort 1B; Cohort 1C; Cohort 1D; Cohort 1E; Cohort 1F; Cohort 2A; Cohort 2B
Drug: leucovorin — 200 (mFOLFOX7) or 400 (mFOLFOX6) mg/m^2 given IV every 2 weeks. Part of FOLFOX regimen.
  Arms: Cohort 1A; Cohort 1B; Cohort 1D; Cohort 1E; Cohort 2A; Cohort 2B
Drug: fluorouracil — 400 mg/m^2 (IV bolus after leucovorin) and/or 2400 mg/m^2 (continuous infusion over 46 hours). Part of FOLFOX regimen.
  Arms: Cohort 1A; Cohort 1B; Cohort 1D; Cohort 1E; Cohort 2A; Cohort 2B
Drug: capecitabine — 1000 mg/m^2 is taken twice per day orally on Days 1-14 of each 3 week cycle. Part of CAPOX regimen.
  Arms: Cohort 1C; Cohort 1F; Cohort 2A
Drug: pembrolizumab — 400 mg given by IV on day 1 of cycle 1, then every 6 weeks.
  Other Names: KEYTRUDA
  Arms: Cohort 1E; Cohort 1F; Cohort 1G; Cohort 2A

SUMMARY:
This trial studies tucatinib to find out if it is safe when given with trastuzumab and other anti-cancer drugs (pembrolizumab, FOLFOX, and CAPOX). It will look at what side effects happen when participants take this combination of drugs. A side effect is anything the drug does other than treating cancer. It will also look at whether tucatinib works with these drugs to treat certain types of cancer.

The participants in this trial have HER2-positive (HER2+) cancer in their gut, stomach, intestines, or gallbladder (gastrointestinal cancer).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an unresectable or metastatic solid malignancy that is histologically or cytologically confirmed to be one of the tumor types listed below:

  * Cohorts 1A, 1B, 1C, and 1D

    * CRC
    * Gastric adenocarcinoma
    * GEJ adenocarcinoma
    * Esophageal adenocarcinoma
    * Cholangiocarcinoma
    * Gallbladder carcinoma
  * Cohorts 1E, 1F, 1G, and 2A

    * Gastric adenocarcinoma
    * GEJ adenocarcinoma
    * Esophageal adenocarcinoma
  * Cohort 2B

    * CRC
* Participants must be candidates to receive an oxaliplatin-based regimen as part of their standard-of-care treatment for all cohorts, except Cohort 1G.
* HER2+ disease, as determined by historic or local laboratory testing
* Phase 1b cohorts: measurable or non-measurable disease according to RECIST v1.1 as determined by the investigator
* Phase 2 cohorts: measurable disease according to RECIST v1.1 as determined by the investigator
* Eastern Cooperative Oncology Group Performance Status score of 0 or 1.

Exclusion Criteria:

* History of known hypersensitivity to planned study treatment
* Known to be positive for Hepatitis B or C
* For Cohorts 2A and 2B: prior anti-HER2 therapies
* For Cohorts 1E, 1F, 1G, 2A: Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE)

There are additional inclusion criteria. The study center will determine if criteria for participations are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (21):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - University of Colorado Denver CTO(CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - PCM Trials, Denver, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Duke University Medical Center, Duke Cancer Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research., Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTUC-024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with unresectable or metastatic human epidermal growth factor receptor 2 positive (HER2+) gastrointestinal (GI) cancer were enrolled across Japan and the United States.
Pre-assignment Details: The study consisted of two phases: phase 1b (dose escalation) consisting of cohorts 1A, 1B, 1D, 1E and 1F and phase 2 (dose expansion) consisting of Cohort 2B. Cohorts 1C and 1G (Phase 1b) and Cohort 2A (Phase 2) were also planned; however, sponsor decided to close the enrollment before these cohorts were opened, therefore no data is reported for Cohorts 1C, 1G and 2A in any section of the results. Data is reported at the primary completion date.
Groups:
- Cohort 1A: Participants received tucatinib 150 milligrams (mg) orally (PO) twice daily (BID) on Days 1 to 14, loading dose of trastuzumab at 6 milligram per kilogram (mg/kg) via intravenous (IV) infusion on Day 1 of Cycle 1 followed by 4 mg/kg once every 2 weeks (Q2W) starting on Cycle 2 Day 1 and mFOLFOX 6 or mFOLFOX7 (oxaliplatin 85 milligram per meter square (mg/m^2) IV, leucovorin 400 mg/m^2 [mFOLFOX6] or 200 mg/m^2 [mFOLFOX7] administered IV, fluorouracil 400 mg/m^2 [IV bolus] [mFOLFOX6] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle. Each cycle was of 14 days. Participants continued on therapy until disease progression (PD), unacceptable toxicity, withdrawal of consent, death, or study closure.
- Cohort 1B: Participants received tucatinib 300 mg PO BID on Days 1 to 14, loading dose of trastuzumab at 6 mg/kg via IV infusion on Day 1 of Cycle 1 followed by 4 mg/kg Q2W starting on Cycle 2 Day 1 and mFOLFOX6 or mFOLFOX7 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 [mFOLFOX6] or 200 mg/m^2 [mFOLFOX7] administered IV, fluorouracil 400 mg/m^2 [IV bolus] [mFOLFOX6] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle. Each cycle was of 14 days. Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
- Cohort 1D: Japanese participants received tucatinib 300 mg PO BID on Days 1 to 14, loading dose of trastuzumab at 6 mg/kg via IV infusion on Day 1 of Cycle 1 followed by 4 mg/kg Q2W starting on Cycle 2 Day 1 and mFOLFOX6 or mFOLFOX7 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 [mFOLFOX6] or 200 mg/m^2 [mFOLFOX7] administered IV, fluorouracil 400 mg/m^2 [IV bolus] [mFOLFOX6] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle. Each cycle was of 14 days. Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
- Cohort 1E: Participants received tucatinib 300 mg PO BID on Days 1 to 14 (Each cycle = 14 Days), trastuzumab every three weeks (Q3W) 8 mg/kg via IV infusion on Day 1 of Cycle 1 and then 6 mg/kg every 3 weeks (Q3W) starting on Day 1 of Cycle 2 (Each cycle = 21 Days), mFOLFOX 6 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 administered IV, fluorouracil 400 mg/m^2 [IV bolus] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle (Each cycle = 14 Days) and pembrolizumab 400 mg IV on Day 1 of Cycle 1 and then every six weeks (Q6W) starting on Day 1 of Cycle2 (Each cycle = 42 days). Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
- Cohort 1F: Participants received tucatinib 300 mg PO BID on Days 1 to 14, trastuzumab 8 mg/kg via IV infusion on Day 1 of Cycle 1 followed by 6 mg/kg Q3W starting on Day 1 of Cycle 2 (Each cycle = 21 days), CAPOX (oxaliplatin 130 mg/m^2 IV on Day 1 and capecitabine 1000mg/m^2 PO BID on evening of Day 1 to morning of Day 15 of Cycle 1 and Day 1 to 14 of each subsequent cycle) (Each cycle = 21 Days) and pembrolizumab 400 mg IV on Day 1 of Cycle 1 and then Q6W starting on Day 1 of Cycle 2. Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
- Cohort 2B: Participants received tucatinib 300 mg PO BID on Days 1 to 14, loading dose of trastuzumab at 8 mg/kg via IV infusion on Day 1 of Cycle 1 followed by 6 mg/kg Q2W starting on Cycle 2 Day 1 and mFOLFOX6 or mFOLFOX7 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 [mFOLFOX6] or 200 mg/m^2 [mFOLFOX7] administered IV, fluorouracil 400 mg/m^2 [IV bolus] [mFOLFOX6] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle. Each cycle was of 14 days. Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
Period: Phase 1: Dose Escalation
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1D | Cohort 1E | Cohort 1F | Cohort 2B
Started | 5 | 11 | 7 | 4 | 8 | 0
Completed | 3 | 4 | 0 | 0 | 0 | 0
Not Completed | 2 | 7 | 7 | 4 | 8 | 0
Not completed — Death | 1 | 4 | 4 | 1 | 6 | 0
Not completed — Participation terminated by sponsor | 0 | 2 | 3 | 2 | 2 | 0
Not completed — Continuing to long term extension phase (LTEP) | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Expansion
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1D | Cohort 1E | Cohort 1F | Cohort 2B
Started | 0 | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Participation terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Continuing to LTEP | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1A: Participants received tucatinib 150 mg PO BID on Days 1 to 14, loading dose of trastuzumab at 6 mg/kg via IV infusion on Day 1 of Cycle 1 followed by 4 mg/kg Q2W starting on Cycle 2 Day 1 and mFOLFOX6 or mFOLFOX7 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 [mFOLFOX6] or 200 mg/m^2 [mFOLFOX7] administered IV, fluorouracil 400 mg/m^2 [IV bolus] [mFOLFOX6] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle. Each cycle was of 14 days. Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A | Cohort 1B | Cohort 1D | Cohort 1E | Cohort 1F | Cohort 2B | Total
Number analyzed (Participants) | 5 | 11 | 7 | 4 | 8 | 5 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.7) | 65.4 (12.9) | 61.6 (11.8) | 65.8 (6.3) | 56.5 (17.3) | 60.6 (8.4) | 60.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 1 | 2 | 3 | 15
  Male | 4 | 8 | 2 | 3 | 6 | 2 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 7 | 2 | 7 | 3 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 5 | 9 | 0 | 2 | 1 | 2 | 19
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic, Latino/a, or of Spanish Origin | 5 | 10 | 7 | 4 | 8 | 5 | 39
  Not reportable | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Renal Dose-Limiting Toxicities (DLTs): Phase 1b (Cohort 1A and 1B)
Description: A renal DLT was defined as an increase in serum cystatin C >1.5* baseline that was not related to pre-renal or post-renal etiologies (including disease progression, dehydration and intercurrent illness) and occurred during the period of treatment with tucatinib in combination with trastuzumab and FOLFOX between the first dose of tucatinib and the end of Cycle 3. Increased serum cystatin C for which there was an alternative clinical explanation (eg, clearly related to an intercurrent illness or disease progression) was not considered renal DLTs.
Time Frame: From first dose of tucatinib until end of Cycle 3 (up to 42 days)
Population: The DLT-evaluable analysis set for cohort 1A and 1B included all participants in cohort 1A or 1B who met one of the following criteria: had a renal DLT or had taken at least 75% of planned oxaliplatin and tucatinib doses per cycle and were followed for at least 2 cycles of study treatment (through the end of Cycle 3 for FOLFOX regimens), inclusive of dose delays.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 3 | 8
Participants | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Phase 1b (Cohort 1E and 1F)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment, end of study date, death date, or data cutoff date, whichever was earlier (maximum of 20.7 months)
Population: The safety analysis set included all participants who were enrolled in the study and received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1E: Participants received tucatinib 300 mg PO BID on Days 1 to 14 (Each cycle = 14 Days), trastuzumab Q3W 8 mg/kg via IV infusion on Day 1 of Cycle 1 and then 6 mg/kg Q3W starting on Day 1 of Cycle 2 (Each cycle = 21 Days), mFOLFOX 6 (oxaliplatin 85 mg/m^2 IV, leucovorin 400 mg/m^2 administered IV, fluorouracil 400 mg/m^2 [IV bolus] and then fluorouracil 2400 mg/m^2 administered IV over 46 hours) on Day 1 of each cycle (Each cycle = 14 Days) and pembrolizumab 400 mg IV on Day 1 of Cycle 1 and then Q6W starting on Day 1 of Cycle2 (Each cycle = 42 days). Participants continued on therapy until PD, unacceptable toxicity, withdrawal of consent, death, or study closure.
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 4 | 8

3. Primary Outcome: Number of Participants With Treatment Related TEAEs: Phase 1b (Cohort 1E and 1F)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment. Treatment related TEAEs were AEs related to any study treatment and relatedness was judged by investigator.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 4 | 8

4. Primary Outcome: Number of Participants With Greater Than or Equal to (>=) Grade 3 TEAEs: Phase 1b (Cohort 1E and 1F)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment. TEAEs were graded according to National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v) 5.0 where grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Number of participants with >= grade 3 TEAEs are reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 4 | 7

5. Primary Outcome: Number of Participants With >= Grade 3 Treatment Related TEAEs: Phase 1b (Cohort 1E and 1F)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment. TEAEs were graded according to NCI-CTCAE v 5.0 where grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Treatment related TEAEs were AEs related to study treatment and relatedness was judged by investigator. Number of participants with >= grade 3 treatment related TEAEs are reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 4 | 7

6. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE): Phase 1b (Cohort 1E and 1F)
Description: An SAE was any untoward medical occurrence at any dose that was fatal; life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was medically significant.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 1 | 6

7. Primary Outcome: Number of Participants With Any Treatment Related SAE: Phase 1b (Cohort 1E and 1F)
Description: An SAE was any untoward medical occurrence at any dose that was fatal; life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was medically significant. Treatment related SAEs were SAEs related to any study treatment and relatedness was judged by investigator.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants | 1 | 5

8. Primary Outcome: Number of Participants With DLTs: Phase 1b (Cohort 1E)
Description: DLTs were AEs/ laboratory abnormalities that were considered to be related to tucatinib/ tucatinib in combination with chemotherapy(mFOLFOX6/CAPOX) and/or trastuzumab and/or pembrolizumab. DLTs was defined any of following: a-)Hepatic- any instance of aspartate aminotransferase(AST)/ alanine aminotransferase(ALT)>3*upper limit of normal(ULN) and total bilirubin >2*ULN that is not thought to be due to progressive disease(PD)/other medical illness. PD:at least 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study. In addition to relative increase of 20%,sum must also demonstrate an absolute increase of at least 5 millimeters(mm). b-) Non-hematologic- any clinically significant, non-hematologic treatment-related AE>= grade(G)3, with following exceptions:G3 fatigue=< 7days,G3 diarrhea,nausea/vomiting without optimal use of anti-emetics/antidiarrheals c-)hematologic:>=G3 febrile neutropenia and absolute neutrophil count(ANC) decreased G4 for >7days.
Time Frame: Cycle 1 (Up to 21 days)
Population: The DLT evaluable analysis set for cohort 1E included all participants who met one of following criteria: had a DLT or had taken at least 75% of planned study treatment for first 21 days of study treatment and were followed for at least 21 days of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E
Number analyzed (Participants) | 3
Participants | 1

9. Primary Outcome: Number of Participants With DLTs: Phase 1b (Cohort 1F)
Description: DLTs were AEs/ laboratory abnormalities that were considered to be related to tucatinib/ tucatinib in combination with chemotherapy (mFOLFOX6/CAPOX) and/ or trastuzumab and/ or pembrolizumab. DLTs was defined any of following: a-) Hepatic- any instance of AST/ ALT >3*ULN and total bilirubin >2*ULN that is not thought to be due to PD/ other medical illness. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. b-) Non-hematologic- any clinically significant, non-hematologic treatment-related AE>= grade 3, with following exceptions: grade 3 fatigue=< 7days, grade 3 diarrhea, nausea/vomiting without optimal use of anti-emetics/antidiarrheals c-) hematologic: >= grade 3 febrile neutropenia and ANC decreased grade 4 for >7days.
Time Frame: Cycle 1 (Up to 28 days)
Population: The DLT evaluable analysis set for cohort 1F included all participants who met one of following criteria: had a DLT or had taken at least 75% of planned study treatment for first 28 days of study treatment and were followed for at least 28 days of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1F
Number analyzed (Participants) | 5
Participants | 0

10. Primary Outcome: Number of Participants With Treatment Emergent Hematological Laboratory Abnormalities: Phase 1b (Cohort 1E and 1F)
Description: The following hematological parameters were assessed: hemoglobin decreased, leukocytes decreased, lymphocytes decreased, neutrophils decreased and platelets decreased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment. Hematological laboratory abnormalities were graded according to NCI CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with hematological abnormalities of any grade were reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants
  Hemoglobin decreased | 2 | 7
  Leukocytes decreased | 4 | 3
  Lymphocytes decreased | 4 | 5
  Neutrophils decreased | 4 | 2
  Platelets decreased | 3 | 8

11. Primary Outcome: Number of Participants With Treatment Emergent Chemistry Laboratory Abnormalities: Phase 1b (Cohort 1E and 1F)
Description: The following chemistry laboratory parameters were assessed: alanine aminotransferase (ALT) increased, albumin decreased, alkaline phosphatase increased, aspartate aminotransferase (AST) increased, calcium corrected for albumin decreased, creatinine increased, calcium corrected for albumin increased, lactate dehydrogenase increased, potassium decreased, potassium increased, sodium decreased, sodium increased and total bilirubin increased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil, oxaliplatin and pembrolizumab) through 30 days after the last dose of study treatment Chemistry laboratory abnormalities were graded according to NCI CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with chemistry abnormalities of any grade were reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants
  ALT increased | 3 | 7
  Albumin decreased | 2 | 5
  Alkaline Phosphatase increased | 0 | 2
  AST increased | 2 | 7
  Calcium Corrected for Albumin decreased | 1 | 4
  Creatinine increased | 1 | 3
  Calcium Corrected for Albumin increased | 0 | 1
  Lactate Dehydrogenase increased | 3 | 3
  Potassium decreased | 4 | 5
  Potassium increased | 1 | 1
  Sodium decreased | 3 | 6
  Sodium increased | 1 | 2
  Total Bilirubin increased | 1 | 2

12. Primary Outcome: Number of Participants With Clinically Significant Post-Baseline Vital Signs: Phase 1b (Cohort 1E and 1F)
Description: Vital signs included temperature, blood pressure, heart rate and respiratory rate. Clinically significant vital signs were defined as: temperature greater than or equal to (>=) 38 degrees Celsius, respiratory rate greater than (>) 20 breaths per minute, systolic blood pressure (SBP) >= 120 millimeter of mercury (mmHg) or diastolic blood pressure (DBP) >= 80 mmHg, SBP >= 140 mmHg or DBP >= 90 mmHg and heart rate > 100 beats per minute (bpm).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Participants
  Temperature >= 38 degrees Celcius | 0 | 0
  Respiratory Rate > 20 breaths per minute | 2 | 2
  SBP >= 120 mmHg or DBP >= 80 mmHg | 4 | 8
  SBP >= 140 mmHg or DBP >= 90 mmHg | 4 | 7
  Heart rate > 100 bpm | 2 | 4

13. Primary Outcome: Number of Participants With TEAEs: Phase 1b (Cohort 1D)
Description: An AE was defined as any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment, end of study date, death date, or data cutoff date, whichever was earlier (maximum of 21 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 7

14. Primary Outcome: Number of Participants With Treatment Related TEAEs: Phase 1b (Cohort 1D)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Treatment related TEAEs were AEs related to study treatment and relatedness was judged by investigator.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 7

15. Primary Outcome: Number of Participants With >= Grade 3 TEAEs: Phase 1b (Cohort 1D)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. TEAEs were graded according to NCI-CTCAE v 5.0 where grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Number of participants with >= grade 3 TEAEs are reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 7

16. Primary Outcome: Number of Participants With >= Grade 3 Treatment Related TEAEs: Phase 1b (Cohort 1D)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. TEAEs were graded according to NCI-CTCAE v 5.0 where grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Treatment related TEAEs were AEs related to study treatment and relatedness was judged by investigator. Number of participants with >= grade 3 treatment related TEAEs are reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 6

17. Primary Outcome: Number of Participants With Any SAE: Phase 1b (Cohort 1D)
Description: as for outcome 6
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 3

18. Primary Outcome: Number of Participants With Any Treatment Related SAE: Phase 1b (Cohort 1D)
Description: as for outcome 7
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 0

19. Primary Outcome: Number of Participants With DLTs: Phase 1b (Cohort 1D)
Description: as for outcome 9
Time Frame: Cycle 1 (Up to 28 days)
Population: The DLT-evaluable analysis set for Cohort 1D included all participants who met one of the following criteria: had a DLT or had taken at least 75% of planned fluorouracil, oxaliplatin, trastuzumab, and tucatinib doses and were followed for at least 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 6
Participants | 1

20. Primary Outcome: Number of Participants With Treatment Emergent Hematological Laboratory Abnormalities: Phase 1b (Cohort 1D)
Description: The following hematological parameters were assessed: hemoglobin decreased, leukocytes decreased, lymphocytes decreased, neutrophils decreased and platelets decreased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Hematological laboratory abnormalities were graded according to NCI CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with hematological abnormalities of any grade were reported.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants
  Hemoglobin decreased | 4
  Leukocytes decreased | 7
  Lymphocytes decreased | 5
  Neutrophils decreased | 6
  Platelets decreased | 6

21. Primary Outcome: Number of Participants With Treatment Emergent Chemistry Laboratory Abnormalities: Phase 1b (Cohort 1D)
Description: The following chemistry parameters were assessed: ALT increased, albumin decreased, alkaline phosphatase increased, AST increased, calcium corrected for albumin decreased, creatinine increased, lactate dehydrogenase increased, potassium decreased, potassium increased, sodium decreased and sodium increased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Chemistry laboratory parameters abnormalities were graded according to NCI CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with chemistry abnormalities of any grade were reported.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants
  ALT increased | 6
  Albumin decreased | 1
  Alkaline Phosphatase increased | 3
  AST increased | 5
  Calcium Corrected for Albumin decreased | 3
  Creatinine increased | 5
  Lactate Dehydrogenase increased | 2
  Potassium decreased | 4
  Potassium increased | 1
  Sodium decreased | 6
  Sodium increased | 1

22. Primary Outcome: Number of Participants With Clinically Significant Post-Baseline Vital Signs: Phase 1b (Cohort 1D)
Description: Vital signs included temperature, blood pressure, heart rate and respiratory rate. Clinically significant vital signs were defined as: temperature >= 38 degrees Celsius, respiratory rate > 20 breaths per minute, SBP >= 120 mmHg or DBP >= 80 mmHg, SBP >= 140 mmHg or DBP >= 90 mmHg and heart rate > 100 beats per minute (bpm).
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants
  Temperature >= 38C | 0
  Respiratory Rate > 20 breaths per minute | 2
  SBP >= 120 mmHg or DBP >= 80 mmHg | 6
  SBP >= 140 mmHg or DBP >= 90 mmHg | 6
  Heart rate > 100 bpm | 2

23. Primary Outcome: Number of Participants With TEAEs Leading to Dose Holds: Phase 1b (Cohort 1D)
Description: An AE was defined as any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Dose hold was considered as dose delay and dose elimination. Number of participants with TEAEs leading to dose holds are reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 6

24. Primary Outcome: Number of Participants With TEAEs Leading to Dose Reductions: Phase 1b (Cohort 1D)
Description: An AE was defined as any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Number of participants with TEAEs leading to dose reductions are reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants | 0

25. Primary Outcome: Number of Participants With TEAEs Leading to Dose Discontinuations: Phase 1b (Cohort 1D)
Description: An AE was defined as any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Number of participants with TEAEs leading to dose discontinuations (i.e. permanent withdrawal of tucatinib, trastuzumab, oxaliplatin, fluorouracil and leucovorin) are reported in this outcome measure.
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1D
Number analyzed (Participants) | 7
Participants
  Tucatinib | 2
  Trastuzumab | 1
  Oxaliplatin | 3
  Fluorouracil | 1
  Leucovorin | 1

26. Primary Outcome: Number of Participants With TEAEs: Phase 2 (Cohort 2B)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment, end of study date, death date, or data cutoff date, whichever was earlier (maximum of 20.9 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 5

27. Primary Outcome: Number of Participants With Treatment Related TEAEs: Phase 2 (Cohort 2B)
Description: as for outcome 14
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 5

28. Primary Outcome: Number of Participants With >= Grade 3 TEAEs: Phase 2 (Cohort 2B)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. TEAEs were graded according to NCI-CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Number of participants with >= grade 3 TEAEs are reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 4

29. Primary Outcome: Number of Participants With >= Grade 3 Treatment Related TEAEs: Phase 2 (Cohort 2B)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. TEAEs were graded according to NCI-CTCAE v 5.0 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Treatment related TEAEs were AEs related to study treatment and relatedness was judged by investigator. Number of participants with >= grade 3 treatment related TEAEs are reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 3

30. Primary Outcome: Number of Participants With Any SAE: Phase 2 (Cohort 2B)
Description: as for outcome 6
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 3

31. Primary Outcome: Number of Participants With Any Treatment Related SAE: Phase 2 (Cohort 2B)
Description: as for outcome 7
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants | 1

32. Primary Outcome: Number of Participants With Treatment Emergent Hematological Laboratory Abnormalities: Phase 2 (Cohort 2B)
Description: Following hematological parameters were assessed: hemoglobin decreased, leukocytes decreased, lymphocytes decreased, neutrophils decreased and platelets decreased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Hematological abnormalities were graded according to NCI CTCAE v 5.0; where, grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening). Participants with hematologic abnormalities of any grade were reported.
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants
  Hemoglobin decreased | 2
  Leukocytes decreased | 3
  Lymphocytes decreased | 2
  Neutrophils decreased | 4
  Platelets decreased | 5

33. Primary Outcome: Number of Participants With Treatment Emergent Chemistry Laboratory Abnormalities: Phase 2 (Cohort 2B)
Description: Following chemistry parameters were assessed: ALT increased, albumin decreased, alkaline phosphatase increased, AST increased, creatinine increased, glomerular filtration rate (GFR) estimated decreased, lactate dehydrogenase increased, potassium decreased, potassium increased, sodium decreased, sodium increased and total bilirubin increased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Chemistry abnormalities were graded according to NCI CTCAE v 5.0; where, grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Participants with chemistry abnormalities of any grade were reported.
Time Frame: as for outcome 26
Population: The safety analysis set included all participants who were enrolled in the study and received any amount of study treatment. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants
  ALT increased | 4
  Albumin decreased | 3
  Alkaline phosphatase increased | 1
  AST increased | 3
  Creatinine increased | 3
  GFR, estimated decreased: number analyzed (Participants) | 2
  GFR, estimated decreased | 1
  Lactate dehydrogenase increased | 1
  Potassium decreased | 3
  Potassium increased | 2
  Sodium decreased | 2
  Sodium increased | 1
  Total bilirubin increased | 1

34. Primary Outcome: Number of Participants With Clinically Significant Post-Baseline Vital Signs: Phase 2 (Cohort 2B)
Description: Vital signs included temperature, blood pressure and heart rate. Clinically significant vital signs were defined as: temperature >= 38 degrees Celsius, respiratory rate > 20 breaths per minute, SBP >= 120 mmHg or DBP >= 80 mmHg, SBP >= 140 mmHg or DBP >= 90 mmHg and heart rate > 100 bpm.
Time Frame: as for outcome 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Participants
  Temperature >= 38 degrees Celsius | 0
  Respiratory Rate > 20 breaths per minute | 1
  SBP >= 120 mmHg or DBP >= 80 mmHg | 5
  SBP >= 140 mmHg or DBP >= 90 mmHg | 4
  Heart rate > 100 bpm | 0

35. Secondary Outcome: Number of Participants With TEAEs: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 13
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment, end of study date, death date, or data cutoff date, whichever was earlier (maximum of 38.2 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 5 | 11

36. Secondary Outcome: Number of Participants With Treatment Related TEAEs: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 14
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 4 | 11

37. Secondary Outcome: Number of Participants With >= Grade 3 TEAEs: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 15
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 2 | 8

38. Secondary Outcome: Number of Participants With >= Grade 3 Treatment Related TEAEs: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 16
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 1 | 6

39. Secondary Outcome: Number of Participants With Any SAE: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 6
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 1 | 5

40. Secondary Outcome: Number of Participants With Any Treatment Related SAE: Phase 1b (Cohort 1A and 1B)
Description: as for outcome 7
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants | 0 | 4

41. Secondary Outcome: Number of Participants With Treatment Emergent Hematological Laboratory Abnormalities: Phase 1b (Cohort 1A and 1B)
Description: Following hematological parameters were assessed: hemoglobin decreased, leukocytes decreased, lymphocytes decreased, neutrophils decreased and platelets decreased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Hematological laboratory abnormalities were graded according to NCI CTCAE v 5.0; where, grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Participants with hematological abnormalities of any grade were reported.
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants
  Hemoglobin decreased | 1 | 5
  Leukocytes decreased | 0 | 9
  Lymphocytes decreased | 0 | 8
  Neutrophils decreased | 0 | 7
  Platelets decreased | 2 | 10

42. Secondary Outcome: Number of Participants With Treatment Emergent Chemistry Laboratory Abnormalities: Phase 1b (Cohort 1A and 1B)
Description: Following chemistry parameters were assessed: ALT increased, albumin decreased, alkaline phosphatase increased, AST increased, calcium corrected for albumin decreased, calcium corrected for albumin increased, creatinine increased, Cystatin C increased, GFR estimated decreased, lactate dehydrogenase increased, potassium decreased, potassium increased, sodium decreased and total bilirubin increased. TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, leucovorin, fluorouracil and oxaliplatin) through 30 days after the last dose of study treatment. Chemistry laboratory abnormalities were graded according to NCI CTCAE v 5.0 grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening. Participants with chemistry abnormalities of any grade were reported.
Time Frame: as for outcome 35
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants
  ALT increased | 3 | 6
  Albumin decreased | 2 | 3
  Alkaline Phosphatase increased | 0 | 3
  AST increased | 1 | 3
  Calcium corrected for albumin decreased | 1 | 4
  Calcium corrected for albumin increased | 0 | 1
  Creatinine increased | 0 | 8
  Cystatin C increased | 2 | 8
  GFR estimated decreased: number analyzed (Participants) | 5 | 9
  GFR estimated decreased | 0 | 6
  Lactate dehydrogenase increased: number analyzed (Participants) | 5 | 10
  Lactate dehydrogenase increased | 1 | 4
  Potassium decreased | 0 | 3
  Potassium increased | 0 | 1
  Sodium decreased | 2 | 2
  Total bilirubin increased | 0 | 2

43. Secondary Outcome: Number of Participants With Clinically Significant Post-Baseline Vital Signs: Phase 1b (Cohort 1A and 1B)
Description: Vital signs included temperature, blood pressure, heart rate and respiratory rate. Clinically significant vital signs were defined as: temperature >= 38 degrees Celsius, respiratory rate > 20 breaths per minute, SBP >= 120 mmHg or DBP >= 80 mmHg, SBP >= 140 mmHg or DBP >= 90 mmHg and heart rate > 100 bpm.
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Participants
  Temperature >= 38 degrees Celsius | 0 | 0
  Respiratory Rate > 20 breaths per min | 0 | 1
  SBP >= 120 mmHg or DBP >= 80 mmHg | 5 | 11
  SBP >= 140 mmHg or DBP >= 90 mmHg | 1 | 9
  Heart rate > 100 bpm | 0 | 3

44. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR): Phase 1b (Cohort 1A and 1B)
Description: GFR value was estimated using serum Cystatin C. Baseline was considered as the most recent non-missing measurement prior to the first dose of any study treatment.
Time Frame: Baseline, Cycle 1 Day 3, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 8 (each cycle=14 days)
Population: The safety analysis set included all participants who were enrolled in the study and received any amount of study treatment. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Milliliter per minute per 1.73 meter^2
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 5 | 11
Milliliter per minute per 1.73 meter^2
  Baseline | 91.1 (19.2) | 87.4 (14.6)
  Change at Cycle 1 Day 3: number analyzed (Participants) | 4 | 10
  Change at Cycle 1 Day 3 | -12.0 (10.4) | -17.3 (7.2)
  Change at Cycle 1 Day 8 | 2.7 (6.5) | 0.2 (11.5)
  Change at Cycle 2 Day 1 | 3.7 (4.6) | 0.0 (13.8)
  Change at Cycle 2 Day 3: number analyzed (Participants) | 5 | 10
  Change at Cycle 2 Day 3 | -19.3 (11.9) | -17.0 (14.7)
  Change at Cycle 2 Day 8: number analyzed (Participants) | 3 | 10
  Change at Cycle 2 Day 8 | -4.9 (4.1) | 0.6 (14.5)

45. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 8 Hours (AUC 0-8h) of Tucatinib at Cycle 1 Day 1: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: Predose, 1 hour intra-dose, end of dose, 1, 2, 4, 6 hours after end of 2 hour oxaliplatin infusion (8 hours) on Day 1 of Cycle 1 and 2
Population: The pharmacokinetic (PK) analysis set included all participants in the safety set from whom at least one PK assessment was reported. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter (ng*h/mL)
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
Nanogram*hours per milliliter (ng*h/mL) | 1130 (108) | 1970 (33.5)

46. Secondary Outcome: Maximum Observed Concentration (Cmax) of Tucatinib: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: as for outcome 45
Population: The PK analysis set included all participants in the safety set from whom at least one PK assessment was reported. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
Nanogram per milliliter (ng/mL) | 197 (105) | 403 (42.7)

47. Secondary Outcome: Observed Trough Concentration in Plasma (Ctrough) of Tucatinib: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: Predose on Day 1 of Cycle 2
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
ng/mL | 106 (113) | 255 (45.2)

48. Secondary Outcome: Time at Which the Maximum Plasma Concentration Occurs (Tmax) of Tucatinib: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: as for outcome 45
Population: as for outcome 46
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
hours | 3.50 [0.950 to 4.20] | 4.08 [1.0 to 7.97]

49. Secondary Outcome: AUC 0-8h of Oxaliplatin: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: as for outcome 45
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter (ng*h/mL)
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
Nanogram*hours per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 10400 (13.5) | 11200 (22.8)
  Cycle 2 Day 1 | 11600 (20.2) | 12100 (10.2)

50. Secondary Outcome: Cmax of Oxaliplatin: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: as for outcome 45
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
Nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 2200 (6.42) | 2240 (15.4)
  Cycle 2 Day 1 | 2250 (15.7) | 2350 (10.9)

51. Secondary Outcome: Tmax of Oxaliplatin: Phase 1b (Cohort 1A and 1B)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: as for outcome 45
Population: as for outcome 46
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 4 | 7
Hours
  Cycle 1 Day 1 | 2.08 [2.03 to 2.13] | 2.12 [2.0 to 2.20]
  Cycle 2 Day 1 | 2.10 [2.0 to 2.27] | 2.03 [1.85 to 2.18]

52. Secondary Outcome: Objective Response Rate (ORR) Per Investigator (INV): Phase 1b (Cohort 1E and 1F)
Description: ORR was defined as percentage of participants with confirmed complete response (CR)/ partial response (PR) per investigator according to response evaluation criteria in solid tumors version 1.1 (RECIST) v1.1. For response to be considered confirmed, subsequent response had to be at least 4 weeks after initial response. CR: complete disappearance of all target lesions with exception of nodal disease and complete disappearance of non-target lesions and normalization of tumor marker level. Any pathological lymph nodes(whether target/ non-target) must have reduction in short axis to <10 mm. PR: >= 30% decrease in sum of diameters of target lesions, taking as reference baseline sum of diameters. 90% exact confidence interval (CI) was based on Clopper-Pearson method.
Time Frame: From the first dose of study treatment until the first documented CR or PR or before start of any new anti-cancer therapy (up to 24.1 months)
Population: The response evaluable set included all participants who met all following criteria: had measurable disease at baseline, received any amount of study treatment, and had at least one post-baseline disease assessment or discontinued due to clinical progression, toxicity or death.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 6
Percentage of Participants | 100.0 [47.3 to 100.0] | 66.7 [27.1 to 93.7]

53. Secondary Outcome: Duration of Response (DOR) Per INV: Phase 1b (Cohort 1E and 1F)
Description: DOR was defined as time from first documented objective response (CR or PR that was subsequently confirmed) to first documented PD per RECIST v1.1 or death due to any cause, whichever occurred first. PD: at least a 20 % increase in sum of diameters of target lesions, taking as reference smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. CR: complete disappearance of all target lesions with exception of nodal disease and complete disappearance of non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: a >= 30 % decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters. 90% exact CI was based on Clopper-Pearson method.
Time Frame: From the first documented objective response until the first documentation of PD or death due to any cause, whichever occurred first (up to 18.1 months)
Population: The response evaluable set included all participants who met all following criteria: had measurable disease at baseline, received any amount of study treatment, and had at least one post-baseline disease assessment or discontinued due to clinical progression, toxicity or death. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for the outcome measure.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 4
Months | 15.5 [4.9 to NA] — Upper limit of 90% CI could not be estimated due to insufficient number of participants with events | 12.4 [4.3 to NA] — Upper limit of 90% CI could not be estimated due to insufficient number of participants with events

54. Secondary Outcome: Progression Free Survival (PFS) Per INV: Phase 1b (Cohort 1E and 1F)
Description: PFS as per INV was defined as time from the date of treatment initiation to date of documented PD as assessed by INV per RECIST version 1.1 or death from any cause, whichever occurred first. Participants without documentation of progression or death at the time of analysis were censored at the date of the last disease assessment. PD: at least 20 % increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered progression.
Time Frame: From the first dose of study treatment until the first documented PD or death from any cause or censoring date, whichever occurred first (up to 24.1 months)
Population: The full analysis set (FAS) included all participants who were enrolled in the study and receive any amount of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 8
Months | 18.3 [2.8 to 19.7] | 5.7 [1.4 to 17.8]

55. Secondary Outcome: Overall Survival (OS): Phase 1b (Cohort 1E and 1F)
Description: OS was defined as the time from treatment initiation to death due to any cause. For a participant who was not known to have died by the end of study follow-up, observation of OS was censored on date the participant was last known to be alive (i.e., the date of last contact). Participants lacking data beyond the day of treatment initiation had their survival time censored on date of treatment initiation.
Time Frame: From date of start of study treatment until date of death or censoring date
Population: The full analysis set included all participants who were enrolled in the study and receive any amount of study treatment.
Reporting Status: Not Posted, anticipated posting 2026-09

56. Secondary Outcome: Ctrough of Tucatinib: Phase 1b (Cohort 1E and 1F)
Description: PK parameters were determined using noncompartmental analysis.
Time Frame: Predose on Day 1 of Cycle 2
Population: The PK analysis set included all participants in the safety set from whom at least one PK assessment was reported. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1E | Cohort 1F
Number analyzed (Participants) | 4 | 5
ng/mL | 199 (147) | 185 (113)

57. Secondary Outcome: Confirmed Objective Response Rate (cORR) Per INV: Phase 2 (Cohort 2B)
Description: cORR was defined as the percentage of participants with a confirmed CR or PR per investigator according to RECIST v1.1. For a response to be considered confirmed, the subsequent response had to be at least 4 weeks after the initial response. CR: complete disappearance of all target lesions with exception of nodal disease and complete disappearance of non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: a >= 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. 90% exact CI was based on Clopper-Pearson method.
Time Frame: From the first dose of study treatment until the first documented CR or PR or before start of any new anti-cancer therapy (up to 20.9 months)
Population: as for outcome 52
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Percentage of participants | 80.0 [34.3 to 99.0]

58. Secondary Outcome: DOR Per INV: Phase 2 (Cohort 2B)
Description: as for outcome 53
Time Frame: From the first documented objective response until the first documentation of PD or death, whichever occurred first (up to 19.9 months)
Population: The response evaluable set included all participants who met all following criteria- had measurable disease at baseline, received any amount of study treatment, and had at least one post-baseline disease assessment or discontinued due to clinical progression, toxicity or death. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for the outcome measure.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 2B
Number analyzed (Participants) | 4
Months | NA [11.2 to NA] — Median and upper limit of 90% CI could not be estimated due to insufficient number of participants with events

59. Secondary Outcome: PFS Per INV: Phase 2 (Cohort 2B)
Description: as for outcome 54
Time Frame: From the first dose of study treatment until the first documented PD or death from any cause or censoring date, whichever occurred first (up to 20.9 months)
Population: The FAS included all participants who were enrolled in the study and receive any amount of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 2B
Number analyzed (Participants) | 5
Months | 13.8 [4.6 to 20.9]

60. Secondary Outcome: OS Per INV: Phase 2 (Cohort 2B)
Description: as for outcome 55
Time Frame: From date of start of study treatment until date of death or censoring date
Population: The FAS included all participants who were enrolled in the study and receive any amount of study treatment.
Reporting Status: Not Posted, anticipated posting 2026-09

ADVERSE EVENTS:
Time Frame: All-cause mortality: maximum up to 38.2 months for cohort 1A, 1B and 1D; 24.1 months for cohort 1E and 1F and 20.9 months for cohort 2B. For Treatment emergent SAEs and non-SAEs- From first dose of study treatment (Day 1) up to 30 days after last dose, end of study date, death date/ data cutoff date, whichever was earlier (maximum of 38.2 months: cohort 1A and 1B; 21 months: cohort 1D; 20.7 months: cohort 1E and1F; 20.9 months: cohort 2B)
Description: Same event may appear as both non-serious adverse event and serious adverse event (SAE); however, are presented as distinct events. Event may be categorized as serious in 1 participant and non-serious in another or may have experienced both SAE and non-SAE. All enrolled analysis set included all participants who were enrolled in the study.
Arm/Group | COHORT 1A | COHORT 1B | COHORT 1D | COHORT 1E | COHORT 1F | COHORT 2B
All-Cause Mortality (participants affected / at risk) | 1/5 | 4/11 | 4/7 | 1/4 | 6/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 5/11 | 3/7 | 1/4 | 6/8 | 3/5
Other Adverse Events (participants affected / at risk) | 5/5 | 11/11 | 7/7 | 4/4 | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1A (N=5) | COHORT 1B (N=11) | COHORT 1D (N=7) | COHORT 1E (N=4) | COHORT 1F (N=8) | COHORT 2B (N=5)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1A (N=5) | COHORT 1B (N=11) | COHORT 1D (N=7) | COHORT 1E (N=4) | COHORT 1F (N=8) | COHORT 2B (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 5 (22) | 2 (2) | 1 (4) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 6 (24) | 4 (10) | 2 (6) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (8) | 3 (21) | 2 (4) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (7) | 4 (4) | 1 (1) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 11 (91) | 5 (6) | 3 (5) | 8 (18) | 5 (11)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (8) | 5 (6) | 3 (4) | 3 (10) | 6 (13) | 2 (4)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pigmentation lip (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 4 (18) | 2 (6) | 2 (2) | 4 (4) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (11) | 1 (1) | 2 (3) | 4 (7) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 9 (14) | 3 (3) | 2 (8) | 2 (2) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (10) | 1 (2)
Temperature intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystatin C increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (8) | 3 (5) | 4 (11) | 5 (6) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (1) | 2 (4) | 1 (1) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (11) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (10) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 5 (7) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 5 (7) | 3 (3) | 1 (1) | 5 (6) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (7) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (9) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 4 (7) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (3) | 2 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04430738/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT04430738/SAP_001.pdf